CLINICAL TRIAL: NCT01190332
Title: Conventional Versus Rendezvous Technique of Intraoperative Endoscopic Retrograde Cholangiopancreatography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: ahmed abdel-raouf el-geidie, gastroenterology surgical center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 7918
Record Dates: First submitted 2010-07-06; First posted 2010-08-27 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-02

CONDITIONS: Common Bile Duct Gallstones
Keywords: common bile duct stones
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- conventional technique of ERCP (Placebo Comparator)
  Interventions: Procedure: endoscopic sphincterotomy by conventional method
- Rendezvous technique (Active Comparator)
  Interventions: Procedure: endoscopic sphincterotomy by rendezvous method

INTERVENTIONS:
Procedure: endoscopic sphincterotomy by conventional method
  Arms: conventional technique of ERCP
Procedure: endoscopic sphincterotomy by rendezvous method
  Arms: Rendezvous technique

SUMMARY:
One of the new methods for management of common bile duct stones is intraoperative endoscopic sphincterotomy. It can be performed by many techniques. In the study the investigators compare two methods to find out the best technique for intraoperative endoscopic sphincterotomy.

ELIGIBILITY:
Inclusion Criteria:

* patients with MRCP evidence of common bile duct stones

Exclusion Criteria:

* cholangitis pancreatitis ASA GRADE III, IV Unfit for laparoscopy unfit for ERCP

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2007-10; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
success/failure rate of common bile duct stones removal

SECONDARY OUTCOMES:
complication rate

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology Surgical Center, Al Mansurah, Dakahlia Governorate, Egypt